CLINICAL TRIAL: NCT02487316
Title: A Multicenter Prospective Study of Treatment ALK(+) Systemic Anaplastic Large Cell Lymphoma With Crizotinib
Brief Title: A Study of Treatment ALK(+) Systemic Anaplastic Large Cell Lymphoma With Crizotinib
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Jun Zhu (Other)
Collaborators: Peking University First Hospital (Other); Peking University People's Hospital (Other); Peking University Third Hospital (Other); Peking Union Medical College Hospital (Other); Beijing Hospital (Other Government); Chinese PLA General Hospital (Other); First Hospitals affiliated to the China PLA General Hospital (Other Government); Air Force General Hospital of the PLA (Other Government); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Anhui Provincial Hospital (Other Government); Zhejiang University (Other)
Responsible Party: Sponsor-Investigator, Jun Zhu, Department of Hematology Oncology, clinical oncology college, Director of department, Party Secretary, Peking University
Organization: Peking University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKU-2015052005
Record Dates: First submitted 2015-06-30; First posted 2015-07-01 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Systemic Anaplastic Large-Cell Lymphoma
Keywords: Anaplastic Large Cell Lymphoma; anaplastic lymphoma kinase rearrangement; crizotinib; CHOP chemotherapy
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic | interventions — Crizotinib; R-CHOP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- crizotinib combined with chemotherapy (Experimental): crizotinib 250mg, bid from day 1 to 18 weeks. cyclophosphamide, 750mg/m2,d1, vincristine, 1.4mg/m2, maximal dose is 2mg d1, doxorubicin, 50mg/m2d1, prednison, 100 mg d1-5) every 3 weeks for up to six cycles.
  Interventions: Drug: crizotinib

INTERVENTIONS:
Drug: crizotinib — crizotinib 250mg, oral, bid from day 1 to 18 weeks. cyclophosphamide, 750mg/m2,d1, vincristine, 1.4mg/m2, maximal dose is 2mg d1, doxorubicin, 50mg/m2d1, prednison, 100 mg d1-5) every 3 weeks for up to six cycles.
  Other Names: CHOP chemotherapy

SUMMARY:
The purpose of this study is to determine the efficacy and safety of crizotinib combined with CHOP chemotherapy for patients with ALK(+) Systemic Anaplastic Large Cell Lymphoma.

DETAILED DESCRIPTION:
ALK(+) Systemic Anaplastic Large Cell Lymphoma patients are treated with crizotinib when they receive CHOP chemotherapy. crizotinib 250mg twice a day is administrated from day 1 of chemotherapy to 18 weeks. standard CHOP chemotherapy (cyclophosphamide, 750mg per square meter of body-surface area,d1, vincristine, 1.4mg per square meter of body-surface area, maximal dose is 2mg d1, doxorubicin, 50mg per square meter of body-surface area d1, plus prednison, 100 mg d1-5) every 3 weeks for up to six cycles.

ELIGIBILITY:
Inclusion Criteria:

* primary ALK(+) systemic anaplastic large cell lymphoma histologically confirmed by biopsy without therapy
* ECOG 0-2
* more than 1 measurable lesions with major axis >1.5cm and minor axis>1.0cm
* estimated survival >/3months
* Age 18-65 years
* Women of childbearing age should have a negative pregnancy test; men and women who need to agree to use effective contraception during the period of treatment and the following 1 years
* Signature of informed consent

Exclusion Criteria:

* Age <\ 18years
* without ALK(+) systemic anaplastic large cell lymphoma histologically confirmed by biopsy
* without measurable lesions
* being treated by other drugs in other clinical trials
* Pregnant or lactating women, who are not willing to take contraceptive measures during the study period, or are not willing to use effective contraceptive measures during the period of treatment and the following 1 years
* Hepatic insufficiency: serum total bilirubin, ALT more than 2 times higher than normal
* Renal insufficiency: more than 2 times higher than that of normal serum creatinine
* Blood screening period: WBC < 1 * 109/L * 109/L; platelet < 25; Hb < 60g/L
* HIV test positive

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | 2 years

SECONDARY OUTCOMES:
disease-free survival | 2 years
overall survival | 2 years
objective response rate | 2 years
incidence of >/Grade 3 non-hematology toxicity adverse events | 2 years
QOL assessment | 2 years
  using a battery of cognitive and quality-of-life (QoL) measures

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, MD, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Weiping Liu, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Boi M, Zucca E, Inghirami G, Bertoni F. Advances in understanding the pathogenesis of systemic anaplastic large cell lymphomas. Br J Haematol. 2015 Mar;168(6):771-83. doi: 10.1111/bjh.13265. Epub 2015 Jan 6. PMID 25559471